CLINICAL TRIAL: NCT02790632
Title: Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Efficacy and Safety Study Comparing EG-1962 to Standard of Care Oral Nimodipine in Adults With Aneurysmal Subarachnoid Hemorrhage
Brief Title: Study of EG-1962 Compared to Standard of Care Oral Nimodipine in Adults With Aneurysmal Subarachnoid Hemorrhage
Acronym: NEWTON2
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: DMC review concluded study has a low probability of meeting its primary endpoint
Sponsor: Edge Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EG-01-1962-03
Record Dates: First submitted 2016-05-26; First posted 2016-06-06 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Subarachnoid Hemorrhage, Aneurysmal
Keywords: Aneurysm, Ruptured; Nimodipine; Subarachnoid Hemorrhage
MeSH Terms: conditions — Subarachnoid Hemorrhage; Aneurysm, Ruptured | interventions — EG-1962

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EG-1962 Group (Experimental): * 1 dose of intraventricular EG-1962 (nimodipine microparticles) 600 mg
  * Up to 21 days of placebo capsules/tablets
  Interventions: Drug: EG-1962 (nimodipine microparticles)
- Enteral Nimodipine Group (Active Comparator): * 1 dose of intraventricular normal saline
  * Up to 21 days of oral nimodipine capsules/tablets
  Interventions: Drug: Enteral Nimodipine

INTERVENTIONS:
Drug: EG-1962 (nimodipine microparticles) — Single intraventricular administration of EG-1962 via EVD and placebo capsules or tablets administered for up to 21 days
  Arms: EG-1962 Group
Drug: Enteral Nimodipine — Enteral Nimodipine capsules or tablets administered for up to 21 days and single intraventricular administration of saline via EVD
  Arms: Enteral Nimodipine Group

SUMMARY:
This study compares EG-1962 to enteral nimodipine in the treatment of aneurysmal subarachnoid hemorrhage.

ELIGIBILITY:
Inclusion Criteria:

1. Ruptured saccular aneurysm confirmed by angiography and repaired by neurosurgical clipping or endovascular coiling
2. External ventricular drain in place
3. Subarachnoid hemorrhage on computed tomography (CT) scan of grade 2-4 on the modified Fisher scale
4. WFNS grade 2, 3, or 4

Exclusion Criteria:

1. Major complication during aneurysm repair such as, but not limited to, massive intraoperative hemorrhage, brain swelling, arterial occlusion or inability to secure the ruptured aneurysm
2. Angiographic vasospasm prior to randomization
3. Evidence of a cerebral infarction with neurological deficit

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 374 (Estimated)
Dates: Start 2016-07; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with a favorable outcome measured on the Extended Glasgow Outcome Scale [Primary Efficacy Endpoint] | 90 Days
  Proportion of subjects with a favorable outcome measured on the Extended Glasgow Outcome Scale (GOSE) at Day 90

SECONDARY OUTCOMES:
Proportion of subjects with favorable neurocognitive outcome measured by the Montreal Cognitive Assessment [Secondary Efficacy Endpoint] | 90 Days
  Proportion of subjects with favorable neurocognitive outcome measured by the Montreal Cognitive Assessment (MoCA) at Day 90

OTHER OUTCOMES:
Adverse Events | 90 Days
  Incidence and severity of adverse events in EG-1962 treated subjects compared to subjects treated with standard of care oral nimodipine
Delayed Cerebral Infarction | 30 Days
  Proportion of subjects with delayed cerebral infarction present on CT scan at Day 30

CONTACTS AND LOCATIONS:
Overall Officials: R. Loch Macdonald, MD, PhD, Study Chair — Edge Therapeutics Inc
Locations (79):
- United States (45):
  - University of Alabama at Birmingham Hospital, Birmingham, Alabama
  - Dignity Health; St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - University of California, San Francisco-Fresno, Fresno, California
  - Keck Hospital of USC, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - UCSF, San Francisco, California
  - Yale New Haven Hospital (YNHH), New Haven, Connecticut
  - UF Health Shands Florida, Gainesville, Florida
  - Baptist Medical Center/Lyerly Neurosurgery, Jacksonville, Florida
  - Mayo Clinic Florida, Jacksonville, Florida
  - Tallahassee Neurological Clinic, Tallahassee, Florida
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Illinois Hospital and Health Sciences System, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kentucky Medical Center, Lexington, Kentucky
  - University of Louisville Hospital, Louisville, Kentucky
  - University of Maryland Medical Systems, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - University of New Mexico Hospital, Albuquerque, New Mexico
  - North Shore University Hospital, Manhasset, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Lenox Hill Hospital, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Montefiore Medical Center, The Bronx, New York
  - UNC Hospitals Neuroscience Intensive Care Unit, Chapel Hill, North Carolina
  - Duke University Medical Pavilion, Durham, North Carolina
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Jefferson Hospital for Neuroscience, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC Presbyterian Hospital, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston Air Force Base, South Carolina
  - Semmes Murphey Neurological Clinic, Memphis, Tennessee
  - Inova Fairfax Medical Campus, Falls Church, Virginia
  - VCU Medical Center, Richmond, Virginia
  - University of Washington, Harborview Medical Center, Seattle, Washington
- Australia (3):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Nepean Hospital, Kingswood, New South Wales
  - Royal Adelaide Hospital, Adelaide
- Medizinische Universitat Innsbruck/Tirol Universitatsklinik fur Neurologie, Innsbruck, Austria
- Canada (5):
  - University of Alberta Hospital/Mackenzie Health Sciences Centre, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - St. Michael's Hospital, Toronto, Ontario
  - Centre Hospitalier de l'Universite de Montreal (CHUM), Hopital Notre Dame, Montreal, Quebec
  - Royal University Hospital, Saskatoon, Saskatchewan
- Czechia (4):
  - Faculty Hospital Hradec Kralove, Hradec Králové, Hradec Kralov
  - Faculty Hospital Brno, Brno, South Moravian
  - Faculty Hospital Ostrava, Ostrava
  - Military University Hospital Prague, Prague
- Finland (2):
  - Tampere University Hospital, Tampere, Pirkanmaa
  - Helsinki University Hospital, Helsinki
- Germany (11):
  - Neuro Intensive Care Unit 102i; Campus Charite Mitte (CCM), Berlin
  - Zentrum fur Neurochirurgie der Uniklinik Koln, Cologne
  - Universitatsklinikum Erlangen, Neurologische Klinik, Koptkliniken, Erlangen
  - Klinik für Neurochirurgie des Universitätsklinikum Essen, Essen
  - Klinik für Neurochirurgie, Zentrum der Neurologie und Neurochirurgie, Goethe-Universitätsklinikum Frankfurt am Main, Frankfurt am Main
  - Universitätsklinikum Hamburg Eppendorf, Klinik und Poliklinik für Neurochirurgie, Neues Klinikum, Hamburg
  - Neurochirurgische Klinik der Universität Heidelberg, Heidelberg
  - Klinik und Poliklinik für Neurochirurgie des Universitatsklinikum Leipzig, Leipzig
  - Neurochirurgische Klinik, Universitatsmedizin Mannheim, Universität Heidelberg, Mannheim
  - Neurochirurgische Klinik und Poliklinik, Klinikum rechts der Isar der Technischen Universitat Munchen, München
  - Neutochirurgische Klinik und Poliklinik des Universitatsklinikum Wurzburg, Würzburg
- Hong Kong (2):
  - Queen Mary Hospital, Hong Kong
  - Prince of Wales Hospital, New Kowloon
- Israel (4):
  - Rabin Medical Center, Petah Tikva, Petah-Tikva
  - Rambam Health Care Center, Haifa
  - Hadassah Hebrew University Medical Center, Jerusalem
  - Sheba Medical Center, Ramat Gan
- Auckland City Hospital, Auckland, New Zealand
- National Neuroscience Institute, Singapore, Singapore

REFERENCES:
- [Derived] Carlson AP, Hanggi D, Wong GK, Etminan N, Mayer SA, Aldrich F, Diringer MN, Schmutzhard E, Faleck HJ, Ng D, Saville BR, Bleck T, Grubb R Jr, Miller M, Suarez JI, Proskin HM, Macdonald RL; NEWTON Investigators. Single-Dose Intraventricular Nimodipine Microparticles Versus Oral Nimodipine for Aneurysmal Subarachnoid Hemorrhage. Stroke. 2020 Apr;51(4):1142-1149. doi: 10.1161/STROKEAHA.119.027396. Epub 2020 Mar 6. PMID 32138631
- [Derived] Hanggi D, Etminan N, Mayer SA, Aldrich EF, Diringer MN, Schmutzhard E, Faleck HJ, Ng D, Saville BR, Macdonald RL; NEWTON Investigators. Clinical Trial Protocol: Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Efficacy, and Safety Study Comparing EG-1962 to Standard of Care Oral Nimodipine in Adults with Aneurysmal Subarachnoid Hemorrhage [NEWTON-2 (Nimodipine Microparticles to Enhance Recovery While Reducing TOxicity After SubarachNoid Hemorrhage)]. Neurocrit Care. 2019 Feb;30(1):88-97. doi: 10.1007/s12028-018-0575-z. PMID 30014184